CLINICAL TRIAL: NCT01195012
Title: Pilot Randomized Controlled Trial for Feasibility of an Obesity "Prevention Plus" Intervention for Primary Care Pediatrics: Helping HAND
Brief Title: Pilot RCT of an Obesity Intervention for Primary Care Pediatrics: Helping HAND
Acronym: Helping HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Teresia O'Connor, Associate Professor, Pediatrics-Nutrition, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Purpose: Other
Other Study IDs: BCM-H-22657
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Childhood Obesity
Keywords: child; primary care; treatment; parenting; lifestyle behaviors
MeSH Terms: conditions — Pediatric Obesity | interventions — Diet, Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wait-list control arm (Other): Participants wait-listed to start the behavioral obesity treatment program (Helping HAND) after time two data collection (7 months after baseline).
  Interventions: Behavioral: Helping HAND (Healthy Nutrition and Activity Directions)
- Intervention arm (Experimental): see intervention description
  Interventions: Behavioral: Helping HAND (Healthy Nutrition and Activity Directions)

INTERVENTIONS:
Behavioral: Helping HAND (Healthy Nutrition and Activity Directions) — 6-month behavioral intervention targeting 5-8 year old children and their parents to improve the child's lifestyle behaviors to improve their weight status. The families met monthly with trained Health Advisors for individual sessions in the pediatric clinic with phone calls in between visits to check on progress.

SUMMARY:
This is a feasibility study to evaluate a 6-month obesity treatment intervention (Helping HAND: Health Activity and Nutrition Directions) for pediatric primary care clinics. The program targets 5-8 year old children and their parents to change the child's lifestyle behaviors and the associated parenting practices to improve the child's weight status. Four community clinics participated. Families were recruited from clinics and after informed consent and baseline data have been obtained, the families were randomized into one of two groups: (1) the treatment group who immediately participated in Helping HAND or (2) the wait list control group, who started the program 7 months later. Data were gathered on all the participating children and their parents at three time points: baseline, post the intervention (month 7) and post the wait list control group completing the intervention (month 14).

This was a pilot study to test the feasibility of an obesity prevention plus program delivered in the child's primary care clinic. The primary outcome was family attendance to the 3 data-collection meetings with research staff and the 6 prevention plus intervention sessions with a trained Health Advisor.

ELIGIBILITY:
Inclusion Criteria:

* 1) Child: Healthy 5 to 8 year old child who is overweight (BMI =/>85%), but not morbidly obese (BMI<99%)
* 2) Child attends one of 4 TCPA clinics
* 3) Child is Texas Children's Health Plan member/participant
* 4) Parent who is child's primary care taker able and willing to participate
* 5) Parent and child willing to attend and participate in 6 month intervention sessions and 3 measurement time points over 14 months
* 6) Only one child per family will be eligible to participate.

Exclusion Criteria:

* 1) Parent unable to read or write in English or Spanish.
* 2) Parent or child unable to participate in counseling sessions in English or Spanish
* 3) Child with BMI =/> 99%tile
* 4) Child with medical consequences of obesity (such as hypertension, hypercholesterolemia, insulin resistance, type 2 diabetes) that would require treatment and not prevention.
* 5) Child on medications (such as oral steroids, stimulants, or anti-psychotic medications) that can affect their weight status
* 6) Child with medical problems that could influence their diet or physical activity or make it difficult for that child to participate in a behavior change program (such as mental retardation, neurologic disorders, severe food allergies or severe cardiac or pulmonary disease that restricts their activities).
* 7) Parents who participated in interviews during the developmental phase of Helping HAND
* 8) Family currently participating in other weight treatment of prevention programs

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] O'Connor TM, Hilmers A, Watson K, Baranowski T, Giardino AP. Feasibility of an obesity intervention for paediatric primary care targeting parenting and children: Helping HAND. Child Care Health Dev. 2013 Jan;39(1):141-9. doi: 10.1111/j.1365-2214.2011.01344.x. Epub 2011 Nov 9. PMID 22066521